CLINICAL TRIAL: NCT03120611
Title: Comparison of Two Exercise Programs Intradialysis: Virtual Reality Exercise Versus Conventional Exercise
Brief Title: Virtual Reality Versus Conventional Exercise Intradialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Collaborators: Hospital de Manises, Valencia (Unknown)
Responsible Party: Principal Investigator, Eva Segura Ortí, Principal investigator, Cardenal Herrera University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/0193
Record Dates: First submitted 2017-04-10; First posted 2017-04-19 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: End Stage Renal Disease
Keywords: Exercise; Hemodialysis; Virtual Reality
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity | interventions — Exergaming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtural reality exercise (Experimental): Virtual reality exercise performed during the hemodialysis session, using the Kinect, specially adapted for patients undertaking hemodialysis
  Interventions: Other: Virtual Reality Exercise
- Conventional exercise intradialysis (Active Comparator): Exercise combining both aerobic (cycling) and strengthening exercise of lower limbs for patients during the hemodialysis session
  Interventions: Other: Conventional exercise intradialysis

INTERVENTIONS:
Other: Virtual Reality Exercise — Game developed by the Kinect, adapted to the lying position of participants.
  Arms: Virtural reality exercise
Other: Conventional exercise intradialysis — Aerobic exercise (cycling) and strengthening exercise for lower limbs using elastic bands and gravity
  Arms: Conventional exercise intradialysis

SUMMARY:
All participants exercised during 16 weeks following a conventional intradialysis exercise program. The last 4 weeks of the study participants were randomized into two different exercise programs intradialysis. One group exercised through a virtual reality exercise adapted specially for patients while receiving hemodialysis treatment. The other group exercised with a conventional exercise program, combining aerobic cycling and strengthening exercises.

DETAILED DESCRIPTION:
The first 16 weeks all participants followed an intradialysis exercise program. The exercise program consisted of strengthening exercises for lower limbs and for the upper limb free of fistula. The exercise program included isotonic exercises for quadriceps, triceps surae, psoas, glutei, and brachial biceps; and isometric exercises for hip adductors and hamstrings. Elastic bands were used to apply resistance. Progression was achieved from increasing from 1 set of 10 repetitions until 3 sets of 15 repetitions. This first part lasted no more than 30 minutes. The program also included aerobic exercise (cycling) for up to 30 minutes. Intensity was adapted through the duration of the study so that the participant felt the exercise from hard to somewhat hard (13 to 15 at the rate of perceived exertion 6 to 20). Time and resistance were adapted progressively.

The last four weeks of the program participants were randomized into virtual reality exercise or conventional exercise group. The virtual reality exercise group undertook 30 minutes of exercise. After warming up, participants had to play to an adapted 'treasure hunt' game. Their legs movements were the players projected into an individual tv that gave them feedback regarding their achievements. The aim of the game was to achieve the higher possible score.They moved to pick up coins and to avoid bombs. An adapted Kinect technology was used for the game development.

ELIGIBILITY:
Inclusion Criteria:

- Patients in HD therapy at least 3 months

Exclusion Criteria:

* recent myocardial infarction (within 6 weeks)
* unstable angina
* malignant arrhythmias
* above the knee amputation without replacement
* cerebral vascular disease (ictus, transient ischemia)
* musculoskeletal and respiratory disorders that can get worse with exercise
* impossibility to achieve functional testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Sit to Stand to Sit test 10 | 20 weeks
  Time required to stand up from a chair and sit down 10 consecutive times

SECONDARY OUTCOMES:
Short Physical Performance Battery | 20 weeks
  Balance, gait speed and sit to stand to sit 5 times
Timed Up and Go | 20 weeks
  Time to stand up, walk a short distance, turn, walk back and sit down to the chair again
One leg stand test | 20 weeks
  Time to keep balance on one leg
Sit to Stand to Sit test 60 seconds | 20 weeks
  Number of repetitions achieved of standing up from a chair during 60 seconds
Handgrip | 20 weeks
  Handgrip strength right and left hands
One leg heel rise test | 20 weeks
  Number of repetitions of standing on toes in both legs
6 minutes walk test | 20 weeks
  Number of meters covered during 6 minutes of walking
Adherence | 20 weeks
  Sessions performed/offered
Physical Activity | 16 weeks
  Human activity profile, adjusted and maximal activity score
Physical Activity | 16 weeks
  Physical activity score for the elderly
Inflammatory markers | 16 weeks
  Interleukin 6 (IL6)
Inflammatory markers | 16 weeks
  Monocyte chemoattractant protein-1 (MCP-1)
Inflammatory markers | 16 weeks
  C-Reactive Protein (CRP)
Inflammatory markers | 16 weeks
  Human Tumor Necrosis Factor α (TNF-α)
Health-related quality of life | 16 weeks
  SF-36 subscales and components
Oxidative stress markers | 16 weeks
  Malondialdehyde (MDA)
Oxidative stress markers | 16 weeks
  Carbonylated proteins

CONTACTS AND LOCATIONS:
Overall Officials: Rafael García Maset, MD, Study Chair — Hospital de Manises
Locations (1):
- Hospital de Manises, Manises, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No